CLINICAL TRIAL: NCT04486391
Title: A Multicenter, Open-Label, Randomized Controlled Phase 3 Study of Tislelizumab Monotherapy Versus Salvage Chemotherapy in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Tislelizumab Monotherapy Versus Salvage Chemotherapy for Relapsed/Refractory Classical Hodgkin Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has voluntarily discontinued due to a change in the company-level development strategy and is not because of any safety concern.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-314; CTR20201517 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab (Experimental): Tislelizumab monotherapy for up to 45 months
  Interventions: Drug: Tislelizumab
- Salvage chemotherapy (Experimental): Salvage chemotherapy for up to 45 months
  Interventions: Drug: Salvage Chemotherapy

INTERVENTIONS:
Drug: Tislelizumab — 200 mg administered via intravenous (IV) infusion once every 3 weeks
  Other Names: BGB-A317
  Arms: Tislelizumab
Drug: Salvage Chemotherapy — Salvage chemotherapy administered as assessed as appropriate by the investigator in accordance with the local guideline, including but not limited to DHAP (dexamethasone, cisplatin, high-dose cytarabine), ESHAP (etoposide, methylprednisolone, high-dose cytarabine and cisplatin), DICE (dexamethasone, ifosfamide, carboplatin, etoposide), ICE (ifosfamide, carboplatin, etoposide), IGEV (ifosfamide, gemcitabine, vinorelbine, prednisone), GVD (gemcitabine, vinorelbine, liposomal doxorubicin), and MINE (etoposide, ifosfamide, mesna, mitoxantrone)
  Arms: Salvage chemotherapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy of tislelizumab in participants with relapsed or refractory classical Hodgkin lymphoma (cHL), as measured by Progression-free Survival (PFS) as assessed by investigator

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed cHL.Must have relapsed or refractory ( cHL and

1. Has failed to achieve a response or progressed after autologous hematopoietic stem cell transplant (ASCT). or
2. Has received at least two prior lines of systemic chemotherapies for cHL and is not an ASCT candidate.

   2. Must have measurable disease 3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

   4. Must have adequate organ functions. 5. Prior chemotherapy, radiotherapy, immunotherapy or investigational therapy used to control cancer including locoregional treatment must have been completed ≥ 4 weeks before the first dose of study drug, and all treatment-related adverse events are stable and have either returned to baseline or Grade 0/1

   Key Exclusion Criteria:
   1. Nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma. Known central nervous system (CNS) lymphoma.
   2. Prior allogeneic hematopoietic stem cell transplant. ASCT or Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) within 100 days of first dose of study drug.
   3. Prior therapies targeting PD-1 or PD-L1.
   4. Prior malignancy within the past 3 years except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.
   5. Participant with active autoimmune disease or history of autoimmune disease with high risk of recurrence.
   6. Serious acute or chronic infection requiring systemic therapy.
   7. Known human immunodeficiency virus (HIV), or serologic status reflecting active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

   NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) by Investigator | Up to 45 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first

SECONDARY OUTCOMES:
Duration of Response (DOR) by Investigator | Up to 45 months
  The time from the date that response criteria are first met to the date that PD is objectively documented or death, whichever occurs first
Overall Response Rate (ORR) by Investigator | Up to 45 months
  The proportion of participants who achieves a best overall response of complete response (CR) or partial response (PR)
Rate of Complete Response (CR) by Investigator | Up to 45 months
  The proportion of participants who achieves a best overall response of CR
Time to Response (TTR) by Investigator | Up to 45 months
  Time from the date of randomization to the time the response criteria are first met
Overall survival (OS) | Up to 45 months
  Defined as the time from the date of randomization to the date of death due to any reason
Number of participants experiencing Adverse Events (AEs) | Up to 45 months
Number of participants experiencing Serious Adverse Events (SAEs) | Up to 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Xia Zhao, MD, Study Director — BeiGene
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/